CLINICAL TRIAL: NCT04265027
Title: An Open Label, Randomised, Two Period, Crossover Study to Assess Bioavailability, Bioequivalence and S COMT Activity Between Two Active Pharmaceutical Ingredient Sources of Opicapone at Two Different Dosage Strengths (50 mg and 25 mg) After Single and Multiple Dose Administrations Under Fasting Conditions in Healthy Volunteers.
Brief Title: Bioavailability and Bioequivalence Between Two Active Pharmaceutical Ingredient (API) Sources of Opicapone (OPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BIA-91067-131
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: Ongentys
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (50 mg Dose) (Experimental): Test IMP: 50 mg BIA 9 1067 and Reference IMP: 50 mg Ongentys. The IMPs were administered fasted (after an overnight fast of at least 8 h) with 240 mL water once daily on Days 1 and Days 3 to 12. Subjects remained fasted and sitting upright for at least 4 h after dose. No fluids (apart from water taken with dose) were allowed from 1 h prior to dosing until 1 h afterwards.
  There were at least 14 days between the last dose of treatment period 1 and the first dose of treatment period 2.
  Interventions: Drug: 50 mg BIA 9 1067; Drug: 50 mg Ongentys
- Group 2 (25 mg Dose) (Experimental): Test IMP: 25 mg BIA9 1067 and Reference IMP: 25 mg Ongentys. The IMPs were administered fasted (after an overnight fast of at least 8 h) with 240 mL water once daily on Days 1 and Days 3 to 12. Subjects remained fasted and sitting upright for at least 4 h after dose. No fluids (apart from water taken with dose) were allowed from 1 h prior to dosing until 1 h afterwards.
  There were at least 14 days between the last dose of treatment period 1 and the first dose of treatment period 2.
  Interventions: Drug: 25 mg BIA9 1067; Drug: 25 mg Ongentys

INTERVENTIONS:
Drug: 50 mg BIA 9 1067 — Hard Capsule; Oral
  Other Names: Test IMP
  Arms: Group 1 (50 mg Dose)
Drug: 25 mg BIA9 1067 — Hard Capsule; Oral
  Other Names: Test IMP
  Arms: Group 2 (25 mg Dose)
Drug: 50 mg Ongentys — Hard Capsule; Oral
  Other Names: Reference IMP
  Arms: Group 1 (50 mg Dose)
Drug: 25 mg Ongentys — Hard Capsule; Oral
  Other Names: Reference IMP
  Arms: Group 2 (25 mg Dose)

SUMMARY:
This study evaluates the bioavailability and bioequivalence between two active pharmaceutical ingredient (API) sources of opicapone (OPC) at two different dosage strengths (50 mg and 25 mg) after single and multiple dose administration under fasting conditions in healthy volunteers and assess soluble catechol O methyltransferase (S-COMT) activity in 2 API sources of OPC at two different dosage strengths (50 mg and 25 mg) after single and multiple dose administration under fasting conditions in healthy volunteers

DETAILED DESCRIPTION:
The current study aims to compare the relative bioavailability and assess the bioequivalence and tolerability of 2 different sources of opicapone from test investigational medicinal product (IMP) (BIA 9 1067) and reference IMP (Ongentys®), at doses of 25 mg and 50 mg. This was an open label, randomised, 2 period, single and multiple dose, crossover, pharmacokinetic (PK), pharmacodynamic (PD) study in 2 groups of healthy male and female subjects.

The study comprised a pre-study screen, followed by 2 treatment periods (1 and 2) and a post-study follow-up.

Screening (Day 28 to Day 2): Screening assessments were carried out between 28 and 2 days before first administration of investigational medicinal product (IMP). Eligible subjects were asked to return for the treatment periods. Continued eligibility was confirmed pre dose during each treatment period.

Treatment Periods (Day 1 to Day 14): Eligible subjects received both of the following IMPs over 2 treatment periods (1 IMP/period). Subjects were dosed in 2 groups.

Each treatment period was approximately 15 days duration, from the morning before dosing (Day 1) until the morning of Day 14. During each treatment period, subjects arrived at the Clinical Unit on Day 1. Each IMP was administered once daily on the mornings of Day 1 (single dose) and Days 3 12 (multiple dose), fasted (after an overnight fast of at least 8 hours [h]) with 240 mL water and subjects were discharged on the morning of Day 14 (48 h post last dose). Safety was also evaluated throughout the study. There were at least 14 days between the last dose of treatment period 1 and the first dose of treatment period 2.

Post Study: Post study assessments were conducted 7 to 14 days after subjects had been discharged from their final treatment period (or if early termination occurred).

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study specific screening procedure was performed;
2. Healthy males and females between 18 and 55 years of age (inclusive);
3. Non smoker or ex smokers for at least 3 months prior to screening;
4. Body mass index (BMI) between 18 and 30 kg/m2, inclusive;
5. No clinically significant (CS) history of allergy / sensitivity to BIA 9 1067/OPC or any of the excipients contained within the IMP(s);
6. Negative tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti HCV Ab) and anti human immunodeficiency virus antibodies (anti HIV 1 and HIV 2) at screening;
7. Negative screen for alcohol, cotinine and drugs of abuse at screening and on admission for each treatment period;
8. Healthy as determined by the Investigator based on medical history, physical examination, vital signs (systolic blood pressure ≥ 90 mmHg and ≤ 140 mmHg, diastolic blood pressure ≥ 50 mmHg and ≤ 90 mmHg) and digital 12 lead ECG (PR Interval ≥ 120 msec and ≤ 220 msec, QRS width ≥ 70 msec and ≤ 120 msec, QT interval corrected for heart rate using Bazett's formula [QTcB] 350 450 msec);
9. Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;

   If male:
10. Male subjects and female partner willing to use 2 effective methods of contraception, i.e., established method of contraception and condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse was in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP;
11. Refrained from donating sperm throughout the study and for 3 months after the last dose of IMP;

    If female:
12. Were of non childbearing potential by reason of surgery or at least 1 year post menopause (i.e., 12 months post last menstrual period), or menopause confirmed by follicle stimulating hormone (FSH) testing;
13. Were of childbearing potential, using an effective non hormonal method of contraception (intrauterine device; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomised male partner, provided that he was the sole partner of that subject) for all the duration of the study and for 3 months after the last dose of IMP;
14. Negative serum pregnancy test at screening and negative urine pregnancy test on admission of each treatment period).

Exclusion Criteria:

Any personal or family history of haemostatic disorder; 2. Consumption of more than 21 units (14 units for female subjects) of alcohol a week (1 unit corresponds to 1 glass of 12% wine [10 cL], 1 glass of 40% whisky [2.5 cL], 1 glass of 12% champagne [10 cL], 1 glass of 18% aperitif drink [7 cL] or 1 glass of 5% beer [25 cL]); 3. Use of nicotine replacement products such as patches, gum and/or electronic cigarettes within 3 months prior to the screening visit; 4. Significant infection or known inflammatory process at screening or admission to each treatment period; 5. Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period; 6. Symptomatic orthostatic hypotension (drop of > 20 mmHg in systolic blood pressure and/or > 10 mmHg in diastolic blood pressure) when moving from supine to standing position, together with other symptoms, e.g., dizziness; 7. Previous use of BIA 9 1067; 8. Use of any investigational drug or participation in any clinical study within 90 days or within 5 t1/2, whichever was longer; 9. Participation in more than 3 clinical trials within the 12 months prior to screening; 10. Donation (450 mL or more) or reception of any blood or blood products within the 3 months prior to screening; 11. Vegans, vegetarians or other dietary restrictions (e.g., restrictions for medical, religious or cultural reasons); 12. Unable to communicate reliably with the Investigator; 13. Unlikely to co operate with the requirements of the study; 14. Use of medicines within 28 days (or 5 t1/2 [whichever was longer]) of initiation of treatment intake i.e., use of any prohibited medications or use of any medicine which, in the opinion of the Investigator, may have affected subject safety or study assessments; 15. Clinically relevant history or presence of respiratory, gastrointestinal, hepatic, renal, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders; 16. Clinically relevant surgical history that could have interfered with the PK of the study medications; 17. No medication was permitted throughout the study, except for medications to treat AEs.

18. An abnormal hepatic function based on an overall assessment by the Investigator regarding medical history, physical examination and laboratory tests of hepatic function (alanine aminotransferase [ALT] > 1 x the upper limit of normal [ULN], aspartate aminotransferase [AST] > 1 x the ULN and total bilirubin > 1.5 x the ULN [confirmed by subsequent repeat testing]), as judged by the Chief Investigator. If a laboratory assessment was outside of the reference range at the local laboratory at the screening visit or at baseline, the assessment could have been repeated once, as soon as possible, and in any case before enrolment to rule out laboratory error; 19. Any clinically relevant findings in the laboratory tests, including any abnormality in the coagulation tests; 20. History of alcoholism or drug abuse; 21. Females pregnant or breastfeeding at screening; 22. Subjects with clinically relevant neurologic or psychiatric illness (including psychotic events like hallucinations); 23. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose galactose malabsorption.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma OPC concentration following a single dose (Cmax) - (ng/mL) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacokinetic parameters for the analysis of Bioequivalence
Area under the plasma concentration versus time curve (AUC) from the time of dosing to the time of last measurable concentration (AUC0-t) - (h*ng/mL) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacokinetic parameters for the analysis of Bioequivalence
AUC extrapolated to infinity (AUC0-inf) - (h*ng/mL) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacokinetic parameters for the analysis of Bioequivalence
Maximum observed plasma OPC concentration at steady state (Cmax,ss) - (ng/mL) | Day 12 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacokinetic parameters for the analysis of Bioequivalence
AUC from the time of dosing to 24 h (dosing interval) at steady state (AUC0 tau) - (h*ng/mL) | Day 12 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacokinetic parameters for the analysis of Bioequivalence

SECONDARY OUTCOMES:
Maximum S COMT inhibition, expressed as a (%) (Emax) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours), Day 12 Day 12 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours)
  pharmacodynamic parameters for analysis of S-COMT
Area under the S COMT % inhibition time curve, from the time of dosing to 24 h (AUEC24 - COMT inhib) - (%.h) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours), Day 12 Day 12 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours
  pharmacodynamic parameters for analysis of S-COMT
Area under the S COMT activity (pmol/mg Hb/h) time curve, from the time of dosing to 24 h (AUEC24 - COMT activ) - ((pmol MN/mg Hb/h).h) | Day 1 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours), Day 12 Day 12 (Pre-dose, 0.5 hours, 1 hours, 2-18 hours
  pharmacodynamic parameters for analysis of S-COMT

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided